CLINICAL TRIAL: NCT01525641
Title: Special Survey on Long-term Drug Use of Mirapex®-LA Tablets in Patients With Parkinson's Disease
Brief Title: Safety and Efficacy of Long-term Daily Use of Mirapex®-LA Tablets in Patients With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.680
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Results first posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patient with Parkinson's Disease
  Interventions: Drug: Mirapex LA

INTERVENTIONS:
Drug: Mirapex LA — Pramipexole Hydrochloride Hydrate

SUMMARY:
Post-marketing surveillance (PMS) to investigate the safety and efficacy of long-term daily use of Mirapex®-LA Tablets in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion criteria:

- Patients with Parkinson's disease who have never been treated with Mirapex LA Tablets before enrolment will be included.

Exclusion criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 600
Sampling Method: Non-Probability Sample
Enrollment: 615 (Actual)
Dates: Start 2012-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (118):
- Japan (118):
  - Boehringer Ingelheim Investigational Site 28, Abiko,Chiba
  - Boehringer Ingelheim Investigational Site 86, Akashi,Hyogo
  - Boehringer Ingelheim Investigational Site 13, Akita,Akita
  - Boehringer Ingelheim Investigational Site 9, Aomori,Aomori
  - Boehringer Ingelheim Investigational Site 2, Asahikawa,Hokkaido
  - Boehringer Ingelheim Investigational Site 36, Bunkyo,Tokyo
  - Boehringer Ingelheim Investigational Site 35, Chuo,Tokyo
  - Boehringer Ingelheim Investigational Site 40, Chuo,Tokyo
  - Boehringer Ingelheim Investigational Site 54, Chuo,Yamanashi
  - Boehringer Ingelheim Investigational Site 6, Date,Hokkaido
  - Boehringer Ingelheim Investigational Site 34, Edogawa,Tokyo
  - Boehringer Ingelheim Investigational Site 32, Fuchu,Tokyo
  - Boehringer Ingelheim Investigational Site 22, Fujioka,Gunma
  - Boehringer Ingelheim Investigational Site 46, Fujisawa,Kanagawa
  - Boehringer Ingelheim Investigational Site 48, Fujisawa,Kanagawa
  - Boehringer Ingelheim Investigational Site 24, Fukaya,Saitama
  - Boehringer Ingelheim Investigational Site 53, Fukui,Fukui
  - Boehringer Ingelheim Investigational Site 105, Fukuoka,Fukuoka
  - Boehringer Ingelheim Investigational Site 106, Fukuoka,Fukuoka
  - Boehringer Ingelheim Investigational Site 109, Fukuoka,Fukuoka
  - Boehringer Ingelheim Investigational Site 16, Fukushima,Fukushima
  - Boehringer Ingelheim Investigational Site 60, Gifu,Gifu
  - Boehringer Ingelheim Investigational Site 44, Hadano,Kanagawa
  - Boehringer Ingelheim Investigational Site 62, Hamamatsu,Shizuoka
  - Boehringer Ingelheim Investigational Site 96, Hiroshima,Hiroshima
  - Boehringer Ingelheim Investigational Site 97, Hiroshima,Hiroshima
  - Boehringer Ingelheim Investigational Site 78, Ibaraki,Osaka
  - Boehringer Ingelheim Investigational Site 29, Ichihara,Chiba
  - Boehringer Ingelheim Investigational Site 68, Ichinomiya,Aichi
  - Boehringer Ingelheim Investigational Site 57, Iida,Nagano
  - Boehringer Ingelheim Investigational Site 108, Iiduka,Fukuoka
  - Boehringer Ingelheim Investigational Site 88, Ikoma,Nara
  - Boehringer Ingelheim Investigational Site 103, Imabari,Ehime
  - Boehringer Ingelheim Investigational Site 17, Iwaki,Fukushima
  - Boehringer Ingelheim Investigational Site 3, Iwamizawa,Hokkaido
  - Boehringer Ingelheim Investigational Site 117, Kirishima,Kagoshima
  - Boehringer Ingelheim Investigational Site 111, Kitakyushu,Fukuoka
  - Boehringer Ingelheim Investigational Site 5, Kitami,Hokkaido
  - Boehringer Ingelheim Investigational Site 55, Kofu,Yamanashi
  - Boehringer Ingelheim Investigational Site 70, Konan,Aichi
  - Boehringer Ingelheim Investigational Site 27, Koshigaya,Saitama
  - Boehringer Ingelheim Investigational Site 114, Kumamoto,Kumamoto
  - Boehringer Ingelheim Investigational Site 107, Kurume,Fukuoka
  - Boehringer Ingelheim Investigational Site 77, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 23, Maebashi,Gunma
  - Boehringer Ingelheim Investigational Site 42, Minato,Tokyo
  - Boehringer Ingelheim Investigational Site 116, Miyakonojo,Miyazaki
  - Boehringer Ingelheim Investigational Site 66, Miyoshi,Aichi
  - Boehringer Ingelheim Investigational Site 10, Morioka,Iwate
  - Boehringer Ingelheim Investigational Site 74, Moriyama,Shiga
  - Boehringer Ingelheim Investigational Site 4, Muroran,Hokkaido
  - Boehringer Ingelheim Investigational Site 56, Nagano,Nagano
  - Boehringer Ingelheim Investigational Site 30, Nagareyama,Chiba
  - Boehringer Ingelheim Investigational Site 113, Nagasaki,Nagasaki
  - Boehringer Ingelheim Investigational Site 65, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 67, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 52, Nanao,Ishikawa
  - Boehringer Ingelheim Investigational Site 104, Nangoku,Kouchi
  - Boehringer Ingelheim Investigational Site 50, Niigata,Niigata
  - Boehringer Ingelheim Investigational Site 85, Nishinomiya,Hyogo
  - Boehringer Ingelheim Investigational Site 72, Obu,Aichi
  - Boehringer Ingelheim Investigational Site 61, Ogaki,Gifu
  - Boehringer Ingelheim Investigational Site 92, Ohta,Shimane
  - Boehringer Ingelheim Investigational Site 115, Oita,Oita
  - Boehringer Ingelheim Investigational Site 93, Okayama,Okayama
  - Boehringer Ingelheim Investigational Site 95, Okayama,Okayama
  - Boehringer Ingelheim Investigational Site 118, Okinawa,Okinawa
  - Boehringer Ingelheim Investigational Site 110, Onojo,Fukuoka
  - Boehringer Ingelheim Investigational Site 80, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 81, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 82, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 38, Ota,Tokyo
  - Boehringer Ingelheim Investigational Site 75, Otsu,Shiga
  - Boehringer Ingelheim Investigational Site 76, Otsu,Shiga
  - Boehringer Ingelheim Investigational Site 18, Ryugasaki,Ibaragi
  - Boehringer Ingelheim Investigational Site 43, Sagamihara,Kanagawa
  - Boehringer Ingelheim Investigational Site 47, Sagamihara,Kanagawa
  - Boehringer Ingelheim Investigational Site 25, Saitama,Saitama
  - Boehringer Ingelheim Investigational Site 26, Saitama,Saitama
  - Boehringer Ingelheim Investigational Site 79, Sakai,Osaka
  - Boehringer Ingelheim Investigational Site 83, Sakai,Osaka
  - Boehringer Ingelheim Investigational Site 102, Sakaide,Kagawa
  - Boehringer Ingelheim Investigational Site 58, Saku,Nagano
  - Boehringer Ingelheim Investigational Site 31, Sakura,Chiba
  - Boehringer Ingelheim Investigational Site 98, Sanyōonoda
  - Boehringer Ingelheim Investigational Site 1, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 7, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 8, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 59, Sekigahara,Gifu
  - Boehringer Ingelheim Investigational Site 11, Sendai,Miyagi
  - Boehringer Ingelheim Investigational Site 12, Sendai,Miyagi
  - Boehringer Ingelheim Investigational Site 33, Setagaya,Tokyo
  - Boehringer Ingelheim Investigational Site 69, Seto,Aichi
  - Boehringer Ingelheim Investigational Site 63, Shimoda,Shizuoka
  - Boehringer Ingelheim Investigational Site 64, Shimoda,Shizuoka
  - Boehringer Ingelheim Investigational Site 99, Shimonoseki,Yamaguchi
  - Boehringer Ingelheim Investigational Site 20, Shimotsuke,Tochigi
  - Boehringer Ingelheim Investigational Site 21, Shimotsuke,Tochigi
  - Boehringer Ingelheim Investigational Site 90, Shingu,Wakayama
  - Boehringer Ingelheim Investigational Site 37, Shinjuku,Tokyo
  - Boehringer Ingelheim Investigational Site 39, Shinjuku,Tokyo
  - Boehringer Ingelheim Investigational Site 41, Shinjuku,Tokyo
  - Boehringer Ingelheim Investigational Site 51, Takaoka,Toyama
  - Boehringer Ingelheim Investigational Site 101, Tokushima,Tokushima
  - Boehringer Ingelheim Investigational Site 112, Tosu,Saga
  - Boehringer Ingelheim Investigational Site 71, Toyokawa,Aichi
  - Boehringer Ingelheim Investigational Site 84, Toyonaka,Osaka
  - Boehringer Ingelheim Investigational Site 87, Toyooka,Hyogo
  - Boehringer Ingelheim Investigational Site 73, Tsu,Mie
  - Boehringer Ingelheim Investigational Site 19, Tsukuba,Ibaragi
  - Boehringer Ingelheim Investigational Site 94, Tsukubo,Okayama
  - Boehringer Ingelheim Investigational Site 15, Tsuruoka,Yamagata
  - Boehringer Ingelheim Investigational Site 89, Wakayama,Wakayama
  - Boehringer Ingelheim Investigational Site 91, Yazu,Tottori
  - Boehringer Ingelheim Investigational Site 45, Yokohama,Kanagawa
  - Boehringer Ingelheim Investigational Site 49, Yokohama,Kanagawa
  - Boehringer Ingelheim Investigational Site 14, Yokote,Akita
  - Boehringer Ingelheim Investigational Site 100, Yoshinogawa,Tokushima

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an Observational study. Patients in the study have received only the standard treatment and no investigational drug was adminstered.
Groups:
- Subjects With Parkinson's Disease (PD): Subjects with Parkinson's Disease (PD) were orally administered Mirapex LA: Pramipexole Hydrochloride Hydrate tablets with starting dose of 0.375 once daily after meal and increased by 0.75 mg/day at week 2. The daily may be increased by 0.75 mg/day at weekly intervals up to maintenance dose (standard dose: 1.5 to 4.5mg/day). subjects with renal impairment were administered with the starting dose of 0.375 every other day for the first week, if necessary the dose may be increased by 0.375mg every week but not exceeding the daily dose of 2.25mg.
Period: Overall Study
Arm/Group | Subjects With Parkinson's Disease (PD)
Started | 615
Completed | 435
Not Completed | 180
Not completed — Case report form not collected | 25
Not completed — No visit since the first visit | 16
Not completed — Adverse Event | 73
Not completed — Lack of Efficacy | 24
Not completed — Improvement | 5
Not completed — Lost to follow-up (relocation) | 1
Not completed — Lost to follow-up (Unknown reason) | 10
Not completed — Lost to follow-up (Changing hospital) | 19
Not completed — Other than stated above | 7

BASELINE CHARACTERISTICS:
Population: Safety set: included all patients who had received treatment with Mirapex®-LA Tablets except those who were found to have no observation after enrolment, invalid registration, or invalid contract.
Arm/Group | Subjects With Parkinson's Disease (PD)
Number analyzed (Participants) | 569
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.87 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 341
  Male | 228

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Adverse Drug Reactions
Description: Percentage of subjects with adverse drug reactions
Time Frame: From baseline up to week 52
Population: Safety set
Measure: Number; unit: percentage of participants
Arm/Group | Subjects With Parkinson's Disease (PD)
Number analyzed (Participants) | 569
percentage of participants | 24.78

2. Secondary Outcome: Clinical Global Impression of Effect
Description: Clinical global impression (CGI) of effect at the last observation, on a rating scale from very much improved to no effect.
Time Frame: Week 52
Population: Efficacy set: included all patients in the "safety set" except those who had no available efficacy data and/or who did not suffer from Parkinsons Disease
Measure: Number; unit: participants
Arm/Group | Subjects With Parkinson's Disease (PD)
Number analyzed (Participants) | 509
participants
  Very much improved | 14
  Much improved | 223
  Minimally improved | 205
  No effect | 67

3. Secondary Outcome: Change From Baseline in Total Score of the UPDRS Part III to Last Observation
Description: Change from baseline at the last observation in the Unified Parkinson's Disease Rating Scale (UPDRS) Part III total score.
  UPDRS Part III (motor examination) measures the extent of physical impairment displayed by the patient. This evaluation consists of 14 separate components of patient's physical status.
  The UPDRS part III score is the sum of the 14 individual components. The UPDRS Part III total score ranges from 0 to 108.A reduction in UPDRS part III score over time corresponds to an improvement in motor activities.
  The following are the 14 separate components:1. Speech 2. Facial expression 3. Tremor at rest 4. Action or postural tremor of hands 5. Rigidity 6. Finger taps 7. Hand movements 8. Rapid alternating movements of hands 9. Leg agility 10. Arising from chair 11. Posture 12. Gait 13. Postural stability 14. Body bradykinesia and hypokinesia.
Time Frame: Baseline and week 52
Population: Efficacy set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subjects With Parkinson's Disease (PD)
Number analyzed (Participants) | 442
units on a scale | -3.73 (8.27)

4. Secondary Outcome: Change From Baseline in the Modified Hoehn & Yahr to Last Observation
Description: Change from baseline at the last observation in the modified Hoehn and Yahr stage. Stages of the Parkinson's disease will be assessed on an 8-degree scale between stage 0 (no sign of the disease) and 5 (wheelchair bound or bedridden unless aided) in steps of 0, 1, 1.5, 2, 2.5, 3, 4 and 5. A reduction in the score over time represents an improvement.
Time Frame: Baseline and week 52
Population: Efficacy set
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Subjects With Parkinson's Disease (PD)
Number analyzed (Participants) | 459
Units on a scale | -0.12 (0.40)

5. Secondary Outcome: Onset or Offset of On and Off Phenomenon in Patients With Concomitant L-DOPA
Description: Number of patients with onset or offset of on-off phenomenon in patients with concomitant levodopa (L-DOPA). On-off phenomenon is the unpredictable shift from mobility - "on" - to a sudden inability to move - "off".
Time Frame: Week 52
Population: Patients in safety set and with concomitant L-DOPA.
Measure: Number; unit: participants
Arm/Group | Subjects With Parkinson's Disease (PD)
Number analyzed (Participants) | 307
participants
  Yes | 43
  No | 262
  Unknown | 2

6. Secondary Outcome: Onset or Offset of Wearing-off Phenomenon in Patients With Concomitant L-DOPA
Description: Number of patients with onset or offset of wearing-off phenomena in patients with concomitant levodopa (L-DOPA). Wearing-off is when Parkinson's symptoms begin to reappear or become noticeably worse before it is time to take the next scheduled dose of medication.
Time Frame: Week 52
Population: Patients in safety set and with concomitant L-DOPA
Measure: Number; unit: participants
Arm/Group | Subjects With Parkinson's Disease (PD)
Number analyzed (Participants) | 307
participants
  Yes | 144
  No | 163

ADVERSE EVENTS:
Time Frame: From baseline upto Week 52.
Arm/Group | Subjects With Parkinson's Disease (PD)
Serious Adverse Events (participants affected / at risk) | 30/569
Other Adverse Events (participants affected / at risk) | 35/569
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects With Parkinson's Disease (PD) (N=569)
Anaemia (Blood and lymphatic system disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastritis erosive (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Gait disturbance (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Bronchopneumonia (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 4
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Posture abnormal (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 2
Dyskinesia (Nervous system disorders) | 2
Parkinson's disease (Nervous system disorders) | 1
Parkinsonism (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 2
Delusion (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects With Parkinson's Disease (PD) (N=569)
Somnolence (Nervous system disorders) | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes